CLINICAL TRIAL: NCT00329693
Title: A Randomised, Double-blind, Parallel Groups, Dose-finding, Placebo-controlled, Multi-centre, Proof of Concept Study Assessing the Effect of 3-wk Treatment With 1 of 3 Oral Doses of Quinagolide & Placebo in Preventing Ovarian Hyperstimulation Syndrome in Women Undergoing Controlled Ovarian Hyperstimulation.
Brief Title: Study Assessing the Effect of 3-week Treatment With One of Three Oral Doses of Quinagolide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FE999051 CS01
Record Dates: First submitted 2006-05-23; First posted 2006-05-25 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Ovarian Hyperstimulation Syndrome
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — quinagolide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Placebo Comparator): Daily Tablets Dosing
  Interventions: Drug: Norprolac
- 2 (Experimental): Daily Tablets Dose
  Interventions: Drug: Norprolac
- 3 (Experimental): Daily Tablets Dosing
  Interventions: Drug: Norprolac
- 4 (Experimental): Daily Tablets Dosing
  Interventions: Drug: Norprolac

INTERVENTIONS:
Drug: Norprolac — Placebo
  Arms: 1
Drug: Norprolac — Quinagolide
  Arms: 2
Drug: Norprolac — Quinagolide
  Arms: 3
Drug: Norprolac — Quinagolide
  Arms: 4

SUMMARY:
Women included in this study are undergoing controlled ovarian hyperstimulation for assisted reproductive technologies (ART) and present with signs of moderate risk of developing OHSS.

DETAILED DESCRIPTION:
No data to be entered.

ELIGIBILITY:
Inclusion Criteria

1. Signed Informed Consent Form, prior to screening evaluations
2. In good physical and mental health
3. Pre-menopausal females between the ages of 21-37 years (both inclusive) at the time of randomisation
4. Infertility for at least 1 year before randomisation, except for proven bilateral tubal infertility

Exclusion Criteria

1. Any clinically significant systemic disease
2. Endocrine or metabolic abnormalities (pituitary, adrenal, pancreas, liver or kidney)
3. History of recurrent miscarriage
4. Undiagnosed vaginal bleeding

Ages: 21 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 182 (Actual)
Dates: Start 2006-06; Primary Completion 2007-08 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
OHSS | 41 days after hCG injection

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (7):
- Spain (7):
  - IVI Barcelona, Ronda General Mitre, 14, Barcelona
  - IVI Bilbao, Paseo Landabarri, 1, Leioa-Bizkaia
  - IVI Madrid, Santiago de Compostela, 88, Madrid
  - IVI Murcia, Navegante Macías del Poyo, 5, Edificio Delfín-Barrio La Flota, Murcia
  - IVI Sevilla, Avda. República Argentina, 58, Seville
  - IVI Valencia, Plaza de la Policía Local, 3, Valencia
  - IVI Vigo, Plaza Francisco Fernández del Riego, 7 (Plaza Elíptica), Vigo (Pontevedra)

REFERENCES:
- [Derived] Tang H, Mourad SM, Wang A, Zhai SD, Hart RJ. Dopamine agonists for preventing ovarian hyperstimulation syndrome. Cochrane Database Syst Rev. 2021 Apr 14;4(4):CD008605. doi: 10.1002/14651858.CD008605.pub4. PMID 33851429
- [Derived] Busso C, Fernandez-Sanchez M, Garcia-Velasco JA, Landeras J, Ballesteros A, Munoz E, Gonzalez S, Simon C, Arce JC, Pellicer A. The non-ergot derived dopamine agonist quinagolide in prevention of early ovarian hyperstimulation syndrome in IVF patients: a randomized, double-blind, placebo-controlled trial. Hum Reprod. 2010 Apr;25(4):995-1004. doi: 10.1093/humrep/deq005. Epub 2010 Feb 6. PMID 20139430